CLINICAL TRIAL: NCT02006173
Title: Safety and Efficacy Study of Hya-Dermis Mixed With Lidocaine Injection for the Improvement of Nasolabial Folds
Brief Title: Safety and Efficacy Study of Lidocaine Mixed Hyaluronate on Nasolabial Folds Correction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: SciVision Biotech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDCT-TAE
Record Dates: First submitted 2013-12-04; First posted 2013-12-10 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Nasolabial Folds Correction; Pain
Keywords: Hya-Dermis mixed with lidocaine on reducing pain
MeSH Terms: conditions — Pain | interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal saline (Placebo Comparator): Participants will be randomly assigned to nasolabial or nasolabial&cheekbone group and receive control treatment (20mg/ml hyaluronic acid mixed with 0.175 ml normal saline) in one side of the face.
  Interventions: Drug: Normal Saline
- Lidocaine (Active Comparator): Participants will be randomly assigned to nasolabial or nasolabial&cheekbone group and receive experiment treatment (20mg/ml hyaluronic acid mixed with 0.175 ml 2% lidocaine) in one side of the face.
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Xylocaine is a 2 % lidocaine hydrochloride contained liquid anesthesia
  Other Names: Xylocaine
  Arms: Lidocaine
Drug: Normal Saline
  Arms: Normal saline

SUMMARY:
This clinical trial is a double-blind, randomized, within-subject controlled, 2-armed, single-center study sponsored by SciVision Biotech Inc. and approved by National Taiwan University Hospital Research Ethics Committee. The aim of this post-marketing study is to evaluate the safety and efficacy of Hya-Dermis mixed with lidocaine, as well as the effectiveness of corrections of Hya-Dermis mixed with lidocaine. Accounting for potential loss to follow-up, the minimum enrollment was statistically determined to be 40 patients.

The study was estimated to be held one and half year including a 0-2 weeks screening period, a day of treatment, and follow-up at month 1, 3, 6, 9, 12. Patient informed consent forms will be obtained before the treatment. A pre-treatment photograph, nasolabial folds (NLF) severity scale scores, and individual aesthetic satisfaction will be the baseline. Two sets of randomized numbers are used, patient numbers and treatment numbers. Participants with odd patient numbers will be assigned to nasolabial group and those with even patient numbers will be assigned to nasolabial&cheekbone group. Participants receive experiment treatment (Hya-Dermis mixed with lidocaine) in one side and control treatment (Hya-Dermis mixed with normal saline) in the other side of the face randomly depending on the treatment numbers. Both physicians and participants are only blind to the treatment assignment. 30 minutes after the injection, a post-photograph will be used to evaluate NLF severity scale scores and global aesthetic improvement scale (GAIS) by physicians. A questionnaire including the Visual Analog Scale (VAS) of pain during the treatment and individual aesthetic satisfaction will be collected from patients. The effectiveness analyses compare NLF severity scale scores and GAIS based on photograph records from physicians, as well as participant questionnaires for each group on every visit. The safety assessment evaluates any recorded adverse events following the device treatment.

ELIGIBILITY:
Inclusion Criteria:

* Be 30 to 60 years of age and of any sex and willing to receive nasolabial folds correction by intradermal injection procedures
* Have ability to understand and comply with the study requirements
* Have approximately symmetrical nasolabial folds with a nasolabial folds severity score of 2-3 and the score difference between two sides is less 1
* Agree to refrain from undergoing other anti-wrinkle treatments in the injective areas 12 months after the injections.
* If female of child-bearing potential, not be breastfeeding, have a negative urine pregnancy test on the treatment day and agree to use any approved contraceptives or medically acceptable method of birth control throughout the study
* Be willing to provide written informed consent prior to any procedures

Exclusion Criteria:

* Have history or active dermal diseases, inflammation, or any related disease, such as infection, psoriasis, and herpes.
* Have history of coagulation defect diseases and still take aspirin, other anti-clotting, or blood activating medications 1 week before the treatments
* Had permanent or semi-permanent implantation on nasolabial areas
* Had dermal-related surgeries history (for example, laser, chemical dermabrasion, fraxel laser, thermocool) 6 months before the treatments.
* Had facial wrinkles and folds corrections (for example, botox or other dermal fillers) 6 months before the study starts
* Have a known history of allergic reactions like hypersensitivity to hyaluronic acid
* Have a known history of allergic reactions to lidocaine other local anesthesia
* Have poor compliance with the study or follow-up schedule

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Pain Visual Analog Scale | 30 miuntes post-treatment
  A quantification of the severity of pain experienced by individuals during the treatments. A scale of 100 mm horizontal line will be labeled by participants to assess pain on both sides of the injected areas 30 minutes after the treatment. The one on the extreme left (0) represents painless while the one on the extreme right (100) is set as the most pain could be imagined by participants.
Adverse events report | From date of treatment to 12 months
  Any adverse events and abnormal physical parameters or reports occurred and disappeared should be monitored throughout the trial. The records should be assessed and keep on track of the severity of individual adverse events and correlation with the treatment.
  Severity assessment:
  To assess the level of severity by rating 0 (none), 1 (mild), 2 (median), and 3 (sever).
  Correlation assessment:
  Physicians evaluate the impact of adverse events for each individual and determine their causality of the treatment. Based on the correlation with the treatment, giving score 0 (no correlated), 1 (low correlated), 2 (suspected correlated), 3 (most likely correlated).
  Adverse events tracking:
  Any adverse events should be reported to the physicians by participants. Physicians keep following up adverse events experienced participants until the event disappeared or the symptoms stabilized.

SECONDARY OUTCOMES:
Nasolabial folds (NLF) severity scale | From the baseline, 30 minutes post-treatment, to every follow-up at 1, 3, 6, 9, 12 months
  Based on Skin Aging Atlas: Volume 2, Asian type photographs13, taking gender and NLF into consideration to quantify the degree of NLF severity. A validated 8-point photographic scale scored the severity grade from 0 (absent) to 7 (extreme) will be used to assess the severity of NLF at baseline, 30 minutes post-treatment, and every follow-up at 1, 3, 6, 9, 12 months.
Global aesthetic improvement scale (GAIS) | 30 minutes post-treatments and follow-ups at 1, 3, 6, 9, 12 months
  To quantify the level of overall aesthetic improvement 30 minutes after treatments and every follow-up at 1, 3, 6, 9, 12 months. A scale from 1 to 5 represent worse (1), no change (2), improved (3), much improved (4), and very much improved (5).
Aesthetic satisfaction questionnaire | From the baseline, 30 minutes post-treatment, to every follow-up at 1, 3, 6, 9, 12 months
  Subjects subjectively assessed overall satisfaction of general appearance toward the effectiveness of the treatment by rating 1 (not at all satisfied), 2 (not satisfied), 3 (neither satisfied nor dissatisfied), 4 (somewhat satisfied), and 5 (highly satisfied).

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Dermatology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Beer K, Beer J. Overview of facial aging. Facial Plast Surg. 2009 Dec;25(5):281-4. doi: 10.1055/s-0029-1243075. Epub 2009 Dec 18. PMID 20024868
- [Background] Sveikata K, Balciuniene I, Tutkuviene J. Factors influencing face aging. Literature review. Stomatologija. 2011;13(4):113-6. PMID 22362337
- [Background] Albert AM, Ricanek K Jr, Patterson E. A review of the literature on the aging adult skull and face: implications for forensic science research and applications. Forensic Sci Int. 2007 Oct 2;172(1):1-9. doi: 10.1016/j.forsciint.2007.03.015. Epub 2007 Apr 16. PMID 17434276
- [Background] Mendelson B, Wong CH. Changes in the facial skeleton with aging: implications and clinical applications in facial rejuvenation. Aesthetic Plast Surg. 2012 Aug;36(4):753-60. doi: 10.1007/s00266-012-9904-3. Epub 2012 May 12. PMID 22580543
- [Background] Romagnoli M, Belmontesi M. Hyaluronic acid-based fillers: theory and practice. Clin Dermatol. 2008 Mar-Apr;26(2):123-59. doi: 10.1016/j.clindermatol.2007.09.001. PMID 18472056
- [Background] van Eijk T, Braun M. A novel method to inject hyaluronic acid: the Fern Pattern Technique. J Drugs Dermatol. 2007 Aug;6(8):805-8. PMID 17763611
- [Background] Colatsky TJ. Mechanisms of action of lidocaine and quinidine on action potential duration in rabbit cardiac Purkinje fibers. An effect on steady state sodium currents? Circ Res. 1982 Jan;50(1):17-27. doi: 10.1161/01.res.50.1.17. No abstract available. PMID 6274542
- [Background] Smith L, Cockerham K. Hyaluronic acid dermal fillers: can adjunctive lidocaine improve patient satisfaction without decreasing efficacy or duration? Patient Prefer Adherence. 2011 Mar 14;5:133-9. doi: 10.2147/PPA.S11251. PMID 21448297
- See also: National Taiwan University Hospital (NTUH) Research Ethics Committee (REC) — http://www.ntuh.gov.tw/en/RECO/default.aspx?PageView=Shared
- See also: Department of Dermatology, National Taiwan University Hospital — http://www.ntuh.gov.tw/en/derm/default.aspx
- See also: Taiwan Food and Drug Administration, Ministry of Health and Welfare — http://www.fda.gov.tw/EN/index.aspx